CLINICAL TRIAL: NCT02137772
Title: A Phase III Randomized, Placebo-controlled Clinical Trial to Evaluate the Safety and Efficacy of MK-8228 (Letermovir) for the Prevention of Clinically Significant Human Cytomegalovirus (CMV) Infection in Adult, CMV-Seropositive Allogeneic Hematopoietic Stem Cell Transplant Recipients
Brief Title: Letermovir (MK-8228) Versus Placebo in the Prevention of Clinically-Significant Cytomegalovirus (CMV) Infection in Adult, CMV-Seropositive Allogeneic Hematopoietic Stem Cell Transplant Recipients (MK-8228-001)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 8228-001; 2013-003831-31 (EudraCT Number); 152923 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Prevention of CMV Infection or Disease
MeSH Terms: conditions — Disease | interventions — letermovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Letermovir (Experimental): Letermovir oral or intravenous (IV) formulation was administered once daily for up to 14 weeks, beginning up to Day 28 days post-transplant. The dose was 240 mg once daily for participants receiving concomitant cyclosporin A and 480 mg once daily for participants not receiving cyclosporin A. Intravenous infusion was administered only to participants who are unable to swallow tablets or who have a condition that may interfere with absorption of the tablets.
  Interventions: Drug: Letermovir
- Placebo (Placebo Comparator): Placebo oral or IV formulation was administered once daily for up to 14 weeks, beginning up to Day 28 post-transplant. The number of placebo tablets was to mimic that for letermovir administration according to the concomitant cyclosporin A status. Intravenous infusion was administered only to participants who are unable to swallow tablets or who have a condition that may interfere with absorption of the tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Letermovir — Letermovir 240 mg / 480 mg tablets, or 240 mg / 480 mg intravenous solution in 250 mL to be infused over 60 minutes.
  Other Names: MK-8228
  Arms: Letermovir
Drug: Placebo — Placebo tablets, or intravenous solution in 250 mL to be infused over 60 minutes.
  Arms: Placebo

SUMMARY:
The study evaluated the efficacy and safety of letermovir (MK-8228) for the prevention of clinically-significant CMV infection in adult, CMV-seropositive recipients of allogeneic hematopoietic stem cell transplant (HSCT). The hypothesis being tested was that MK-8228 is superior to placebo in the prevention of clinically-significant CMV infection through Week 24 post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Has documented seropositivity for CMV within 1 year before hematopoietic stem cell transplant (HSCT)
* Receiving first allogeneic HSCT (bone marrow, peripheral blood stem cell, or cord blood transplant)
* Female or male participant who is not of reproductive potential, or, if of reproductive potential, agrees to true abstinence or to use (or have their partner use) 2 acceptable methods of birth control from the time of consent through 90 days after the last dose of study drug
* Able to read, understand, and complete questionnaires and diaries

Exclusion Criteria:

* Received a previous allogeneic HSCT (previous autologous HSCT is acceptable)
* History of CMV end-organ disease within 6 months before randomization
* Has evidence of CMV viremia (if tested) at any time from either signing of the Informed Consent Form or the HSCT procedure, whichever is earlier, until the time of randomization.
* Received the following within 7 days before screening or plans to receive during the study: ganciclovir, valganciclovir, foscarnet, acyclovir, valacyclovir, or famciclovir
* Received the following within 30 days before screening or plan to receive during the study: cidofovir, CMV hyper-immune globulin, any investigational CMV antiviral agent or biological therapy
* Has suspected or known hypersensitivity to ingredients of MK-8228 (letermovir) formulations
* Has severe hepatic insufficiency within 5 days before randomization
* Has end-stage renal impairment
* Has an uncontrolled infection on the day of randomization
* Requires mechanical ventilation or is hemodynamically unstable at the time of randomization
* Has documented positive results for human immunodeficiency virus (HIV) antibody, hepatitis C virus (HCV) antibody with detectable HCV ribonucleic acid, or hepatitis B surface antigen (HBsAg) within 90 days before randomization
* Has active solid tumor malignancies with the exception of localized basal cell or squamous cell skin cancer or the condition under treatment (for example, lymphoma)
* Is pregnant or expecting to conceive, is breastfeeding, or plans to breastfeed from the time of consent through 90 days after the last dose of study drug
* Is expecting to donate eggs or sperm from the time of consent through 90 days after the last dose of study drug
* Has participated in a study with an unapproved investigational compound (monoclonal antibodies are excepted) or device within 28 days of the first dose of study drug
* Has previously participated in a MK-8228 (letermovir) study
* Has, is, or is planning (during the study) to participate in any study involving administration of a CMV vaccine or another CMV investigational agent
* Is a user of recreational or illicit drugs or has a recent history (<=1 year) of drug or alcohol abuse or dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2014-06-06 (Actual); Primary Completion 2016-08-08 (Actual); Study Completion 2016-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Prohn M, Cho CR, Viberg A, Dykstra K, Davis C, Sabato P, Stone J, Badshah C, Murata Y, Leavitt R, Fancourt C, Macha S. Exposure-Response Analyses of Letermovir Following Oral and Intravenous Administration in Allogeneic Hematopoietic Cell Transplantation Recipients. Clin Pharmacol Ther. 2022 Feb;111(2):485-495. doi: 10.1002/cpt.2456. Epub 2021 Nov 29. PMID 34674258
- [Derived] Prohn M, Viberg A, Zhang D, Dykstra K, Davis C, Macha S, Sabato P, de Alwis D, Iwamoto M, Fancourt C, Cho CR. Population pharmacokinetics of letermovir following oral and intravenous administration in healthy participants and allogeneic hematopoietic cell transplantation recipients. CPT Pharmacometrics Syst Pharmacol. 2021 Mar;10(3):255-267. doi: 10.1002/psp4.12593. Epub 2021 Mar 12. PMID 33440077
- [Derived] Ljungman P, Schmitt M, Marty FM, Maertens J, Chemaly RF, Kartsonis NA, Butterton JR, Wan H, Teal VL, Sarratt K, Murata Y, Leavitt RY, Badshah C. A Mortality Analysis of Letermovir Prophylaxis for Cytomegalovirus (CMV) in CMV-seropositive Recipients of Allogeneic Hematopoietic Cell Transplantation. Clin Infect Dis. 2020 Apr 10;70(8):1525-1533. doi: 10.1093/cid/ciz490. PMID 31179485
- [Derived] Marty FM, Ljungman P, Chemaly RF, Maertens J, Dadwal SS, Duarte RF, Haider S, Ullmann AJ, Katayama Y, Brown J, Mullane KM, Boeckh M, Blumberg EA, Einsele H, Snydman DR, Kanda Y, DiNubile MJ, Teal VL, Wan H, Murata Y, Kartsonis NA, Leavitt RY, Badshah C. Letermovir Prophylaxis for Cytomegalovirus in Hematopoietic-Cell Transplantation. N Engl J Med. 2017 Dec 21;377(25):2433-2444. doi: 10.1056/NEJMoa1706640. Epub 2017 Dec 6. PMID 29211658

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 738 participants were screened, 570 were randomized 2:1 letermovir:placebo, and 565 received at least one dose of study medication.
Pre-assignment Details: Screening could occur up to 15 days before Hematopoietic Stem Cell Transplant (HSCT) and no more than Day 28 post-transplant. From the time of screening to randomization, participants were tested weekly for Cytomegalovirus (CMV) viremia; a positive test resulted in exclusion from the study.
Groups:
- Letermovir: Letermovir oral or intravenous (IV) formulation was administered once daily for up to 14 weeks, beginning up to Day 28 post-transplant. The dose was 240 mg once daily for participants receiving concomitant cyclosporin A and 480 mg once daily for participants not receiving cyclosporin A. Intravenous infusion was administered only to participants who are unable to swallow tablets or who have a condition that may interfere with absorption of the tablets.
Period: Overall Study
Arm/Group | Letermovir | Placebo
Started | 376 (Randomized participants) | 194 (Randomized participants)
Treated Participants | 373 | 192
Completed | 244 | 119
Not Completed | 132 | 75
Not completed — Adverse Event | 6 | 3
Not completed — Death | 71 | 44
Not completed — Lost to Follow-up | 8 | 4
Not completed — Physician Decision | 15 | 5
Not completed — Withdrawal by Subject | 28 | 17
Not completed — Non-compliance with study drug | 1 | 0
Not completed — Not treated | 3 | 2

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Letermovir | Placebo | Total
Number analyzed (Participants) | 376 | 194 | 570
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.8 (13.4) | 50.8 (14.8) | 50.8 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 77 | 239
  Male | 214 | 117 | 331
Risk Stratum for CMV Reactivation [Number; unit: Participants] — High risk: Participants meeting one or more of the following criteria at randomization: 1) Human leukocyte antigen (HLA)-related (sibling) donor with at least one mismatch at an HLA-A, -B or -DR gene loci 2) Haploidentical donor, 3) Unrelated donor with at least one mismatch at HLA- HLA-A, -B, -C or -DRB1 gene loci 4) Use of umbilical cord blood as stem cell source, 5) Use of ex vivo T-cell-depleted grafts, 6) Grade 2 or greater graft-versus-host disease requiring the use of systemic corticosteroids. Low risk: All other participants
  Participants
    High risk | 122 | 54 | 176
    Low risk | 254 | 140 | 394

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinically-significant CMV Infection up to Week 24 Post-transplant
Description: Clinically-significant CMV infection was defined as either one of the following: 1) onset of CMV end-organ disease, or 2) initiation of anti-CMV pre-emptive therapy based on documented CMV viremia and the clinical condition of the participant. The percentage of participants with clinically-significant CMV infection was assessed.
Time Frame: Up to Week 24 post-transplant
Population: The Full Analysis Set (FAS) was all randomized participants who received ≥1 dose of study drug and had no detectable CMV DNA on Day 1 (randomization). Participants who prematurely discontinued or had a missing outcome through the 24-week visit window were considered treatment failure (i.e. Non-completers equal failure [NC=F] approach was used).
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 325 | 170
Percentage of participants | 37.5 | 60.6
Statistical Analysis 1: Comparison: Letermovir vs Placebo; Test type: Superiority or Other; p < 0.0001, Mantel Haenszel — A 1-sided p-value ≤0.0249 for the risk difference was used for declaring statistical significance; The Mantel Haenszel analysis was adjusted for sample size for each stratum (high or low risk for CMV reactivation); Risk Difference (RD) = -23.5, 95% CI 2-sided [-32.5 to -14.6]

2. Secondary Outcome: Time to Onset of Clinically-significant CMV Infection (Kaplan-Meier Estimate of Percentage of Participants With a Qualifying Event at Week 24 Post-transplant)
Description: Clinically-significant CMV infection was defined as either one of the following: 1) onset of CMV end-organ disease, or 2) initiation of anti-CMV pre-emptive therapy based on documented CMV viremia and the clinical condition of the participant. Time to onset of clinically-significant CMV infection was defined from the day of transplantation to the day the participant developed clinically-significant CMV infection, and was analyzed by the Kaplan-Meier method. Participants were censored at the last assessment for participants who discontinued or did not develop clinically-significant CMV infection.
Time Frame: Up to Week 24 post-transplant
Population: All randomized participants who received at least one dose of study drug and had no detectable CMV viral DNA on the day treatment was initiated.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 325 | 170
Percentage of participants | 18.9 [14.4 to 23.5] | 44.3 [36.4 to 52.1]
Statistical Analysis 1: Comparison: Letermovir vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank — Nominal 2-sided p-value; The log rank test was adjusted for sample size for each stratum (high or low risk for CMV reactivation)

3. Secondary Outcome: Percentage of Participants With Clinically-significant CMV Infection up to Week 14 Post-transplant
Description: as for outcome 1
Time Frame: Up to Week 14 post-transplant
Population: The FAS was all randomized participants who received ≥1 dose of study drug and had no detectable CMV DNA on Day 1. Participants who prematurely discontinued or had a missing outcome through the 14-week visit window were considered treatment failure (i.e. NC=F approach was used).
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 325 | 170
Percentage of participants | 19.1 | 50.0
Statistical Analysis 1: Comparison: Letermovir vs Placebo; Test type: Superiority or Other; p < 0.0001, Mantel Haenszel — Nominal 1-sided p-value; The Mantel Haenszel analysis was adjusted for sample size for each stratum (high or low risk for CMV reactivation); Risk Difference (RD) = -31.3, 95% CI 2-sided [-39.9 to -22.6]

4. Secondary Outcome: Percentage of Participants With CMV End-organ Disease up to Week 24 Post-transplant
Description: CMV end-organ disease met per-protocol diagnostic criteria for CMV-pneumonia, gastrointestinal disease, hepatitis, central nervous system disease, retinitis, nephritis, cystitis, myocarditis, pancreatitis, or other disease categories. Only Clinical Adjudication Committee-confirmed CMV end-organ disease was included in this analysis. The percentage of participants with CMV end-organ disease was assessed.
Time Frame: Up to Week 24 post-transplant
Population: The FAS was all randomized participants who received ≥1 dose of study drug and had no detectable CMV DNA on Day 1. A participant with a missing value up to Week 24 was excluded from the analysis (i.e., Data as observed [DAO] approach was used).
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 254 | 123
Percentage of participants | 2.0 | 2.4
Statistical Analysis 1: Comparison: Letermovir vs Placebo; Test type: Superiority or Other; p = 0.4056, Mantel Haenszel — Nominal 1-sided p-value; The Mantel Haenszel analysis was adjusted for sample size for each stratum (high or low risk for CMV reactivation); Risk Difference (RD) = -0.4, 95% CI 2-sided [-4.0 to 3.2]

5. Secondary Outcome: Percentage of Participants With CMV End-organ Disease up to Week 14 Post-transplant
Description: as for outcome 4
Time Frame: Up to Week 14 post-transplant
Population: The FAS was all randomized participants who received ≥1 dose of study drug and had no detectable CMV DNA on Day 1. A participant with a missing value up to Week 14 was excluded from the analysis (i.e., Data as observed [DAO] approach was used).
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 285 | 145
Percentage of participants | 0.4 | 1.4
Statistical Analysis 1: Comparison: Letermovir vs Placebo; Test type: Superiority or Other; p = 0.2258, Mantel Haenszel — Nominal 1-sided p-value; The Mantel Haenszel analysis was adjusted for sample size for each stratum (high or low risk for CMV reactivation); Risk Difference (RD) = -1.0, 95% CI 2-sided [-3.5 to 1.5]

6. Secondary Outcome: Percentage of Participants With Pre-emptive Therapy for CMV Viremia up to Week 14 Post-transplant
Description: Initiation of anti-CMV pre-emptive therapy was based on documented CMV viremia and the clinical condition of the participant. The percentage of participants with initiation of anti-CMV pre-emptive anti-CMV therapy was assessed.
Time Frame: Up to Week 14 post-transplant
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 325 | 170
Percentage of participants | 18.8 | 49.4
Statistical Analysis 1: Comparison: Letermovir vs Placebo; Test type: Superiority or Other; p < 0.0001, Mantel Haenszel — Nominal 1-sided p-value; The Mantel Haenszel analysis was adjusted for sample size for each stratum (high or low risk for CMV reactivation); Risk Difference (RD) = -31.0, 95% CI 2-sided [-39.6 to -22.4]

7. Secondary Outcome: Percentage of Participants With Pre-emptive Therapy for CMV Viremia up to Week 24 Post-transplant
Description: as for outcome 6
Time Frame: Up to Week 24 post-transplant
Population: The FAS was all randomized participants who received ≥1 dose of study drug and had no detectable CMV DNA on Day 1. Participants who prematurely discontinued or had a missing outcome through the 24-week visit window were considered treatment failure (i.e. NC=F approach was used).
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 325 | 170
Percentage of participants | 36.6 | 59.4
Statistical Analysis 1: Comparison: Letermovir vs Placebo; Test type: Superiority or Other; p < 0.0001, Mantel Haenszel — Nominal 1-sided p-value; The Mantel Haenszel analysis was adjusted for sample size for each stratum (high or low risk for CMV reactivation); Risk Difference (RD) = -23.3, 95% CI 2-sided [-32.3 to -14.3]

8. Secondary Outcome: Time to Initiation of Pre-emptive Therapy for CMV Viremia (Kaplan-Meier Estimate of Percentage of Participants With a Qualifying Event at Week 24 Post-transplant)
Description: The need for anti-CMV pre-emptive therapy was based on documented CMV viremia and the clinical condition of the participant. The outcome was calculated from the day of transplantation to the start of anti-CMV pre-emptive therapy, and was analyzed by the Kaplan-Meier method. Participants were censored at the last assessment for participants who discontinued or did not initiate pre-emptive therapy.
Time Frame: Up to Week 24 post-transplant
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 325 | 170
Percentage of participants | 17.2 [12.8 to 21.6] | 42.4 [34.7 to 50.2]
Statistical Analysis 1: Comparison: Letermovir vs Placebo; Test type: Superiority or Other; p < 0.0001, Log Rank — Nominal 2-sided p-value; The log rank test analysis was adjusted for sample size for each stratum (high or low risk for CMV reactivation)

9. Other Pre Specified Outcome: Percentage of Participants With One or More Adverse Events up to Week 48 Post-transplant
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event.
Time Frame: Up to Week 48 post-transplant
Population: All randomized participants who received at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 373 | 192
Percentage of participants | 98.4 | 100.0

10. Other Pre Specified Outcome: Percentage of Participants Discontinued From Study Medication Due to an Adverse Event
Description: as for outcome 9
Time Frame: Up to Week 14 post-transplant
Population: All randomized participants who received at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Letermovir | Placebo
Number analyzed (Participants) | 373 | 192
Percentage of participants | 19.6 | 51.6

ADVERSE EVENTS:
Time Frame: Up to Week 48 post-transplant
Arm/Group | Letermovir | Placebo
Serious Adverse Events (participants affected / at risk) | 202/373 | 115/192
Other Adverse Events (participants affected / at risk) | 360/373 | 186/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letermovir (N=373) | Placebo (N=192)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (10) | 3 (3)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (2) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Chest pain (General disorders) | 1 (2) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1)
Mucosal inflammation (General disorders) | 2 (2) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 4 (4)
Pyrexia (General disorders) | 10 (12) | 4 (4)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Venoocclusive liver disease (Hepatobiliary disorders) | 2 (2) | 3 (3)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Graft versus host disease (Immune system disorders) | 45 (49) | 29 (31)
Transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Adenoviral haemorrhagic cystitis (Infections and infestations) | 0 (0) | 1 (1)
Aspergillus infection (Infections and infestations) | 1 (1) | 2 (2)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
BK virus infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 4 (4) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0)
Cellulitis orbital (Infections and infestations) | 1 (2) | 0 (0)
Cerebral toxoplasmosis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 3 (3) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 2 (2)
Cystitis viral (Infections and infestations) | 1 (1) | 2 (2)
Cytomegalovirus infection (Infections and infestations) | 14 (15) | 15 (15)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Epstein-Barr viraemia (Infections and infestations) | 1 (1) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 3 (3) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fusarium infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis adenovirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Implant site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Meningoencephalitis herpetic (Infections and infestations) | 1 (1) | 1 (1)
Meningoencephalitis viral (Infections and infestations) | 0 (0) | 1 (1)
Mucormycosis (Infections and infestations) | 1 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 15 (15) | 6 (6)
Pneumonia adenoviral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (1)
Retinitis viral (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 8 (8) | 4 (4)
Septic shock (Infections and infestations) | 5 (5) | 7 (7)
Sinusitis (Infections and infestations) | 4 (4) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 4 (4) | 2 (2)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Systemic candida (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)
Viraemia (Infections and infestations) | 3 (3) | 3 (3)
Viral haemorrhagic cystitis (Infections and infestations) | 3 (3) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Delayed engraftment (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transplant failure (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Lactose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tetany (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 4 (4)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23 (23) | 17 (17)
B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Mantle cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mycosis fungoides recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Natural killer-cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Primary myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Neurotoxicity (Nervous system disorders) | 2 (2) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 2 (2)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 7 (7) | 9 (11)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 3 (3) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diffuse alveolar damage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venoocclusive disease (Vascular disorders) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letermovir (N=373) | Placebo (N=192)
Anaemia (Blood and lymphatic system disorders) | 24 (39) | 12 (13)
Febrile neutropenia (Blood and lymphatic system disorders) | 28 (28) | 19 (20)
Neutropenia (Blood and lymphatic system disorders) | 18 (20) | 11 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 27 (32) | 13 (13)
Dry eye (Eye disorders) | 24 (24) | 12 (12)
Abdominal pain (Gastrointestinal disorders) | 49 (53) | 19 (21)
Abdominal pain upper (Gastrointestinal disorders) | 23 (30) | 17 (20)
Constipation (Gastrointestinal disorders) | 30 (30) | 22 (24)
Diarrhoea (Gastrointestinal disorders) | 108 (139) | 51 (64)
Dry mouth (Gastrointestinal disorders) | 21 (22) | 11 (11)
Dyspepsia (Gastrointestinal disorders) | 21 (22) | 6 (8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 11 (11)
Nausea (Gastrointestinal disorders) | 106 (141) | 53 (64)
Stomatitis (Gastrointestinal disorders) | 24 (25) | 14 (14)
Vomiting (Gastrointestinal disorders) | 79 (93) | 35 (40)
Asthenia (General disorders) | 29 (36) | 9 (13)
Chest pain (General disorders) | 20 (21) | 5 (5)
Fatigue (General disorders) | 55 (63) | 26 (30)
Mucosal inflammation (General disorders) | 45 (47) | 24 (24)
Oedema peripheral (General disorders) | 60 (74) | 23 (27)
Pyrexia (General disorders) | 85 (112) | 50 (60)
Graft versus host disease (Immune system disorders) | 147 (173) | 74 (91)
Bacteraemia (Infections and infestations) | 21 (24) | 4 (5)
Cytomegalovirus infection (Infections and infestations) | 55 (65) | 77 (93)
Nasopharyngitis (Infections and infestations) | 19 (22) | 8 (8)
Viraemia (Infections and infestations) | 12 (12) | 12 (12)
Alanine aminotransferase increased (Investigations) | 26 (31) | 17 (20)
Aspartate aminotransferase increased (Investigations) | 21 (24) | 13 (16)
Blood creatinine increased (Investigations) | 39 (43) | 14 (17)
Decreased appetite (Metabolism and nutrition disorders) | 43 (48) | 26 (26)
Hyperglycaemia (Metabolism and nutrition disorders) | 31 (31) | 13 (14)
Hyperkalaemia (Metabolism and nutrition disorders) | 28 (29) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 23 (25) | 12 (13)
Hypomagnesaemia (Metabolism and nutrition disorders) | 24 (24) | 15 (16)
Hyponatraemia (Metabolism and nutrition disorders) | 23 (24) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (31) | 15 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 24 (26) | 20 (22)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 (13) | 10 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 21 (21) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 (24) | 16 (17)
Dizziness (Nervous system disorders) | 29 (30) | 16 (16)
Dysgeusia (Nervous system disorders) | 19 (19) | 10 (10)
Headache (Nervous system disorders) | 58 (68) | 24 (26)
Tremor (Nervous system disorders) | 29 (30) | 13 (14)
Anxiety (Psychiatric disorders) | 23 (23) | 5 (5)
Insomnia (Psychiatric disorders) | 35 (37) | 12 (12)
Acute kidney injury (Renal and urinary disorders) | 35 (37) | 22 (25)
Dysuria (Renal and urinary disorders) | 17 (17) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 62 (70) | 27 (28)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 36 (38) | 9 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 25 (29) | 13 (13)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 32 (34) | 19 (20)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 10 (11)
Dry skin (Skin and subcutaneous tissue disorders) | 31 (32) | 16 (19)
Erythema (Skin and subcutaneous tissue disorders) | 34 (37) | 12 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 31 (35) | 12 (14)
Rash (Skin and subcutaneous tissue disorders) | 90 (109) | 51 (62)
Hypertension (Vascular disorders) | 34 (38) | 23 (24)
Hypotension (Vascular disorders) | 16 (16) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.